CLINICAL TRIAL: NCT04185766
Title: Use of Oral 40% Destrogel to Prevent Hypoglycaemia in Late-term Births and SGA or LGA Term Newborns
Brief Title: Prevention of Hypoglycaemia by Oral 40% Destrogel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Principal Investigator, Giuseppe De Bernando, Principal Investigator, Fondazione Poliambulanza Istituto Ospedaliero
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3286
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Hypoglycaemia Neonatal
Keywords: Prevention; newborn; oral destrogel; hypoglycaemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucose; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (0,5 ml/Kg) (Placebo Comparator)
  Interventions: Dietary Supplement: Administration of a placebo solution (0.5 ml / kg)
- Placebo (1 ml/Kg) (Placebo Comparator)
  Interventions: Dietary Supplement: Administration of a placebo solution (1 ml / kg)
- Destrogel (0,5 ml/Kg) (Experimental)
  Interventions: Dietary Supplement: Administration of 40% glucose in gel (0.5 ml / Kg)
- Destrogel (1 ml/Kg) (Experimental)
  Interventions: Dietary Supplement: Administration of 40% glucose in gel 1 ml / Kg)

INTERVENTIONS:
Dietary Supplement: Administration of a placebo solution (0.5 ml / kg) — 43 newborns at risk of hypoglycaemia to which a placebo solution will be administered (0.5 ml / kg)
  Other Names: Placebo
  Arms: Placebo (0,5 ml/Kg)
Dietary Supplement: Administration of a placebo solution (1 ml / kg) — 43 newborns at risk of hypoglycaemia to which a placebo solution will be administered (1 ml / kg)
  Other Names: Placebo
  Arms: Placebo (1 ml/Kg)
Dietary Supplement: Administration of 40% glucose in gel (0.5 ml / Kg) — 43 newborns at risk of hypoglycaemia to which a solution of dextrose 40% in gel will be administered (0.5 ml / Kg)
  Arms: Destrogel (0,5 ml/Kg)
Dietary Supplement: Administration of 40% glucose in gel 1 ml / Kg) — 43 newborns at risk of hypoglycaemia to which a solution of dextrose 40% in gel will be administered (1 ml / Kg).
  Arms: Destrogel (1 ml/Kg)

SUMMARY:
Neonatal hypoglycemia understood as a reduction in plasma glucose can result in long-term neurological damage. Serious monitoring of neonatal blood glucose is indicated in patients at risk of hypoglycemia. Glycaemic monitoring in the newborn at risk should be started not before of the two hours of life, in fact at birth the neonatal blood glucose values are very low because they are conditioned by the metabolic activity of the foetus in the intrauterine phase, while later these values rise again until arrive at similar values to the adult within 48-72 hours. In recent years, various research groups have been evaluating the possibility of arriving at non-pharmacological prophylaxis of hypoglycemia. In particular, the Hegarty group has set up a protocol that uses dextrose gel at 40% in the risk categories that could reduce the number of hypoglycemia cases and consequently of painful procedures. In 2013 Harris et al. conducted a study to evaluate the failure rate in the treatment of hypoglycaemia in a sample of 242 newborns assigned in the 1:1 ratio to case or control group. The cases were treated with 40% dextrose in gel with a concentration of 200 mg/kg while the controls with a placebo solution. Newborns of both groups were encouraged to feed but if the feeding was insufficient, it was administered breast milk or formula milk through a syringe. Treated group showed a failure rate in reversion of lower hypoglycaemia compared to controls (14% vs 24%, RR = 0.57 (0.33-0.98), p = 0.04). Hegarty et al conducted a clinical trial in which 416 newborns were randomized and assigned to one of 4 types of treatment: dextrose 40% in gel in a single-dose (200 mg/kg) or double-dose (400 mg/kg ) 1 hour after birth or followed by 3 additional doses of dextrose (200 mg/kg) in the first 12 hours. Blood glucose was measured at 2 hours from birth then every 2-4 hours for the first 12 hours of life. The incidence of hypoglycaemia was lower in the treated than in the control group treated with a placebo solution (41% vs 52%, RR = 0.79 (0.64-0.98), p = 0.03). The group of newborns treated with a single administration of gel at a concentration of 200 mg/kg showed a greater reduction in the incidence of hypoglycaemia compared to the other types of treatment (38% vs 56%, RR = 0.66 (0.47-0.99), p=0.04)

DETAILED DESCRIPTION:
Neonatal hypoglycemia understood as a reduction in plasma glucose can result in long-term neurological damage. Hypoglycemia is one of the most frequent metabolic alterations of the newborn. About 30% of all newborns are at risk of hypoglycemia. The neonatal population at risk is mainly children of diabetic mothers, born prematurely, late preterm (34-36,6 weeks of gestational age), born at term (37-42 weeks of gestational age) with low body weight for gestational age ( SGA, <10o percentile) or with high body weight for gestational age (LGA, >90o percentile). The 50% of these infants have hypoglycemia in the first 48 years. It is still controversial today to assign the threshold value below which it is possible to define a condition of neonatal hypoglycemia. In 2011, the American Academy of Pediatrics provided practical guidance for screening and subsequent management of neonatal hypoglycemia in infants at risk. The chosen threshold was 45 mg/dl but they also stated that few studies have shown that the asymptomatic hypoglycaemia condition protracted for a few hours is associated with long-term neurological damage. Studies showing the correlation between plasma blood sugar concentration and long-term neurological adverse events were also influenced by the variable definition of hypoglycemia, the duration of hypoglycemia, the lack of studies case-control and sample size. The other chosen threshold to diagnose hypoglycemia was 47 mg/dl, however without rigorous scientific evidence. Subsequently in 2015 and 2017, two scientific evidence showed that maintaining blood sugar values above 47 mg/dl in the first 48 hours of life in infants at risk of hypoglycemia and in follow-up, did not associate with an increase in incidence of neurosensory type of alteration, at the age of 2 and 4.5 years of life respectively. Furthermore, these papers established the conditions of severe hypoglycemia for plasma glucose values <36 mg/dl and of recurrent hypoglycemia if at least three hypoglycemia episodes were recorded (<47 mg/dl). The pathophysiological mechanisms underlying neonatal hypoglycemia were: the reduced glycogen storage in the liver of the preterm newborn, the reduced availability of amino acids for gluconeogenesis and the inadequate lipid storage as a source of fatty acids that are more evident in preterm. Regarding the causes of persistent hypoglycemia, specified as a hypoglycemia that persists more than 48 hours of life, we must consider: the inappropriate insulin secretion, hypopituitarism, cortisol deficiency, growth hormone deficiency, congenital errors of glucose metabolism, glycogen and fatty acids. Neonatal hypoglycemia can be completely asymptomatic or can manifest with neurogenic/adrenergic signs and symptoms characterized by: sweating, pallor, cyanosis, temperature instability, irritability, starvation, tremors, tachycardia, emesis and neuroglycopenic signs and symptoms characterized by: apnea, hypotonia, hypovalid suction, seizures, up to the come and the exitus.

Serious monitoring of neonatal blood glucose is indicated in patients at risk of hypoglycemia. Glycemic monitoring in the newborn at risk should be started not before of the two hours of life, in fact it is seen that at birth the neonatal blood glucose values are very low because they are conditioned by the metabolic activity of the fetus in the intrauterine phase, while later these values rise again until arrive at similar values to the adult within 48-72 hours. Monitoring is performed by glucometer, capillary EGA or blood sampling performed in patients at risk of painful stress. In recent years, various research groups have been evaluating the possibility of arriving at non-pharmacological prophylaxis of hypoglycemia. In particular, the Hegarty group has set up a protocol that uses dextrose gel at 40% in the risk categories that could reduce the number of hypoglycemia cases and consequently of painful procedures. Body temperature and the state of metabolic and/or respiratory acidosis are among the main factors that influence blood sugar levels in the first 48 hours of life. There are currently no strategies to prevent hypoglycemia. The treatment, in cases of asymptomatic hypoglycemia, is an early administration of milk in formula while in cases of symptomatic hypoglycemia infusion of 10% intravenous glucose is foreseen or early feeding by treatment with breast milk or in formula. However, the administration of milk formulated in the first hours of life causes a reduction in breastfeeding. In severe cases with glycaemia <36 mg/dl, it is practiced intravenous infusion of 10% glucose or dextrose. The 40% dextrose in gel administered orally can be a valid preventive measure in all newborns at risk of hypoglycemia, sons of a diabetic mother, SGA and LGA and improve the probability of successful breast attachment. Dextrose 40% in gel is administered by massaging it into the buccal mucosa to have an optimal effect.

In 2013 Harris et al. conducted a study to evaluate the failure rate in the treatment of hypoglycaemia in a sample of 242 newborns assigned in the 1:1 ratio to case or control group. The cases were treated with 40% dextrose in gel with a concentration of 200 mg/kg while the controls with a placebo solution. Newborns of both groups were encouraged to feed but if the feeding was insufficient it was administered breast milk or formula milk through a syringe. Blood glucose was detected 30 minutes after gel administration but if hypoglycaemia was persistent, it was administered up to 6 doses of gel during the 48 hours of life. Treated group showed a failure rate in reversion of lower hypoglycaemia compared to controls (14% vs 24%, RR = 0.57 (0.33-0.98), p = 0.04). In 2016 Weston et al. reviewed the scientific literature with the aim of evaluating the efficacy of 40% dextrose in gel in preventing hypoglycaemia and in reducing the long-term damage associated with neurodevelopment. Two trials including 312 infants were included. It was found that the administration of the gel reduced the mother-child separation (RR = 0.54, 95% CI = 0.31-0.93) and the probability of exclusive breastfeeding after discharge was increased (RR 1.10, 95% CI from 1.01 to 1.18).

No side effects related to gel administration were detected by investigators, and the group of gel-treated infants showed an increase in blood glucose of 7.2 mg/dl compared to the placebo group. Hegarty et al conducted a clinical trial in which 416 newborns were randomized and assigned to one of 4 types of treatment: dextrose 40% in gel in a single-dose (200 mg/kg) or double-dose (400 mg/kg ) 1 hour after birth or followed by 3 additional doses of dextrose (200 mg/kg) in the first 12 hours. Blood glucose was measured at 2 hours from birth then every 2-4 hours for the first 12 hours of life. The incidence of hypoglycemia was lower in the treated than in the control group treated with a placebo solution (41% vs 52%, RR = 0.79 (0.64-0.98), p = 0.03). The group of newborns treated with a single administration of gel at a concentration of 200 mg/kg showed a greater reduction in the incidence of hypoglycemia compared to the other types of treatment (38% vs 56%, RR = 0.66 (0.47-0.99), p=0.04). Treatment with 40% dextrose in gel also led to a reduction in admissions to NICU due to hypoglycemia compared to the control group (2% vs 13%, RR = 0.12 (0.02-0.90), p = 0.04) and to the number of newborns treated with milk in formula (Mean Difference = -6.00 (-11.58-0.41), p=0.036). Scientific Safety Evidence: No side effects related to the use of 40% dextrose in gel were recorded in all the studies performed. In 2015, the guidelines published by the University of Auckland, New Zealand, stated that the use of dextrose in gel does not change the incidence of neurosensitive disability at 2 years of correct age, moreover, events like crisis convulsive or dead have not been described after the administration of this gel. Moreover, from the analysis of the literature by various scientific search engines including Pubmed, Scholar and others, using as keywords: newborn, hypoglycemia and dextrose gel, until the moment of writing this synopsis, no work has been detected as far as regards the side effects in the use of dextrose gel.

ELIGIBILITY:
Inclusion Criteria

Mothers:

* Favourable for breastfeeding
* BMI between 19-24

Newborns:

* Late preterm (gestational age: 34-36 weeks)
* Term neonates (gestational age: 37-42 weeks), with body weight <10th centile (SGA) or> 90 ° centile according to Bertino's neonatal anthropometric evaluation
* Born from eutocic childbirth
* Rooming-in
* Body temperature between 36.5-37.5 ° C 2.

Exclusion criteria

Mothers:

* Lack of informed consent
* Diabetic mother
* Taking medicines during pregnancy (beta blockers, tolbutamide)

Newborns:

* Major congenital malformations
* Blood sugar <47 mg / dl
* Body temperature <36.5 ° C or> 37.5 ° C
* NICU admissions
* Milk intake in formula
* Intravenous infusion of 10% glucose solution
* Metabolic and respiratory acidosis (pH: 7.28 - 7.38)

Ages: 34 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Change of the incidence of hypoglycaemia in late term newborns and in SGA and LGA term infants | From birth up to 48 hours of life
  To assess whether a single administration of Destrogel 40% micronutrient can reduce the incidence of hypoglycaemia in late term newborns and in SGA and LGA term infants (gestational age: 37-42 weeks).

SECONDARY OUTCOMES:
Change of the incidence of the use of formula milk and the intravenous administration of 10% glucose solution in late term infants and in SGA and LGA term newborns | From birth up to 48 hours of life
  To evaluate whether the administration of the 40% micronutrient Destrogel is able to decrease the incidence of the use of formula milk and the intravenous administration of 10% glucose solution in late term infants and in SGA and LGA term newborns (gestational age: 37-42 weeks), reducing artificial breastfeeding in favour of breastfeeding and also reducing the pain of the newborn during the execution of peripheral venous access for the administration of hypoglycaemia therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Bernardo, MD, Principal Investigator — Poliambulanza Foundation Hospital Institute; Rosario Ippolito, MD, Study Chair — Physician in specialist training of the University of Pavia; Maurizio Giordano, B.Sc., Study Director — Federico II University
Locations (1):
- Poliambulanza Foundation Hospital Institute, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raylene P. The sacred hour: uninterrupted skin-to-skin contact immediately after birth. Newborn & Infant Nursing Reviews 2013; 13:67-72
- [Background] Rana A, Amr M, Patty W, Sandy I, Mandy. Validation Study of: The Effect of Delayed Newborn Bath and Oral Dextrose Gel for Neonatal Hypoglycemia on Improving In-Hospital Exclusive Breastfeeding Rates. Biomed J Sci &Tech Res 4(4) 2018.BJSTR.MS.ID.0001090
- [Background] Oral Dextrose Gel to Treat Neonatal Hypoglycaemia: New Zealand Clinical Practice Guidelines 2015. Department of Paediatrics: Child and Youth Health, University of Auckland, Auckland, New Zealand
- [Result] Thompson-Branch A, Havranek T. Neonatal Hypoglycemia. Pediatr Rev. 2017 Apr;38(4):147-157. doi: 10.1542/pir.2016-0063. PMID 28364046
- [Result] McKinlay CJ, Alsweiler JM, Ansell JM, Anstice NS, Chase JG, Gamble GD, Harris DL, Jacobs RJ, Jiang Y, Paudel N, Signal M, Thompson B, Wouldes TA, Yu TY, Harding JE; CHYLD Study Group. Neonatal Glycemia and Neurodevelopmental Outcomes at 2 Years. N Engl J Med. 2015 Oct 15;373(16):1507-18. doi: 10.1056/NEJMoa1504909. PMID 26465984
- [Result] Engle WA, Kominiarek MA. Late preterm infants, early term infants, and timing of elective deliveries. Clin Perinatol. 2008 Jun;35(2):325-41, vi. doi: 10.1016/j.clp.2008.03.003. PMID 18456072
- [Result] Committee on Fetus and Newborn; Adamkin DH. Postnatal glucose homeostasis in late-preterm and term infants. Pediatrics. 2011 Mar;127(3):575-9. doi: 10.1542/peds.2010-3851. Epub 2011 Feb 28. PMID 21357346
- [Result] McKinlay CJD, Alsweiler JM, Anstice NS, Burakevych N, Chakraborty A, Chase JG, Gamble GD, Harris DL, Jacobs RJ, Jiang Y, Paudel N, San Diego RJ, Thompson B, Wouldes TA, Harding JE; Children With Hypoglycemia and Their Later Development (CHYLD) Study Team. Association of Neonatal Glycemia With Neurodevelopmental Outcomes at 4.5 Years. JAMA Pediatr. 2017 Oct 1;171(10):972-983. doi: 10.1001/jamapediatrics.2017.1579. PMID 28783802
- [Result] Lago P, Frigo AC, Baraldi E, Pozzato R, Courtois E, Rambaud J, Anand KJ, Carbajal R. Sedation and analgesia practices at Italian neonatal intensive care units: results from the EUROPAIN study. Ital J Pediatr. 2017 Mar 7;43(1):26. doi: 10.1186/s13052-017-0343-2. PMID 28270167
- [Result] Hegarty JE, Harding JE, Gamble GD, Crowther CA, Edlin R, Alsweiler JM. Prophylactic Oral Dextrose Gel for Newborn Babies at Risk of Neonatal Hypoglycaemia: A Randomised Controlled Dose-Finding Trial (the Pre-hPOD Study). PLoS Med. 2016 Oct 25;13(10):e1002155. doi: 10.1371/journal.pmed.1002155. eCollection 2016 Oct. PMID 27780197
- [Result] Futatani T, Shimao A, Ina S, Higashiyama H, Fujita S, Ueno K, Igarashi N, Hatasaki K. Capillary Blood Ketone Levels as an Indicator of Inadequate Breast Milk Intake in the Early Neonatal Period. J Pediatr. 2017 Dec;191:76-81. doi: 10.1016/j.jpeds.2017.08.080. PMID 29173326
- [Result] Spatz DL. Helping Mothers Reach Personal Breastfeeding Goals. Nurs Clin North Am. 2018 Jun;53(2):253-261. doi: 10.1016/j.cnur.2018.01.011. PMID 29779517
- [Result] Chertok IR, Raz I, Shoham I, Haddad H, Wiznitzer A. Effects of early breastfeeding on neonatal glucose levels of term infants born to women with gestational diabetes. J Hum Nutr Diet. 2009 Apr;22(2):166-9. doi: 10.1111/j.1365-277X.2008.00921.x. Epub 2009 Feb 13. PMID 19226355
- [Result] Barber RL, Ekin AE, Sivakumar P, Howard K, O'Sullivan TA. Glucose Gel as a Potential Alternative Treatment to Infant Formula for Neonatal Hypoglycaemia in Australia. Int J Environ Res Public Health. 2018 Apr 27;15(5):876. doi: 10.3390/ijerph15050876. PMID 29702618
- [Result] Weston PJ, Harris DL, Battin M, Brown J, Hegarty JE, Harding JE. Oral dextrose gel for the treatment of hypoglycaemia in newborn infants. Cochrane Database Syst Rev. 2016 May 4;(5):CD011027. doi: 10.1002/14651858.CD011027.pub2. PMID 27142842
- [Result] Harris DL, Weston PJ, Signal M, Chase JG, Harding JE. Dextrose gel for neonatal hypoglycaemia (the Sugar Babies Study): a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Dec 21;382(9910):2077-83. doi: 10.1016/S0140-6736(13)61645-1. Epub 2013 Sep 25. PMID 24075361

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT04185766/Prot_SAP_000.pdf